CLINICAL TRIAL: NCT06780826
Title: A Simulated RCT Study on the Efficacy of Atezolizumab Combined with Chemotherapy Versus Placebo Combined with Chemotherapy in Small Cell Lung Cancer
Brief Title: A Study on the Efficacy of Atezolizumab Combined with Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of the Clinical Research Center, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: SHDC2024CRI067
Record Dates: First submitted 2024-12-12; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer, Small Cell
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Etoposide; Carboplatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- atezolizumab combined with chemotherapy: Patients receive atezolizumab in combination with carboplatin and etoposide
  Interventions: Drug: Atezolizumab; Drug: Etoposide; Drug: Carboplatin
- chemotherapy: Patients received carboplatin and etoposide
  Interventions: Drug: Etoposide; Drug: Carboplatin

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab, 1200 mg intravenous infusion, 21 days per cycle
  Other Names: Tecentriq
  Groups: atezolizumab combined with chemotherapy
Drug: Etoposide — Etoposide,intravenous infusion, 100mg/m,21 days per cycle
  Other Names: VP16
Drug: Carboplatin — carboplatin,intravenous infusion, AUC=5, 21 days per cycle.
  Other Names: CBP

SUMMARY:
This is a multicenter phase III simulated RCT study aimed to compare the efficacy and safety of atezolizumab combined with chemotherapy versus placebo combined with chemotherapy in small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Male or female, 18 years of age or older
* ECOG performance status of 0 or 1
* Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group (VALG) staging system
* No prior treatment for ES-SCLC
* Patients with a history of treated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

  1. Only supratentorial and cerebellar metastases allowed (i.e., no metastases
  2. to midbrain, pons, medulla or spinal cord)
  3. No ongoing requirement for corticosteroids as therapy for CNS disease
  4. No stereotactic radiation within 7 days
  5. No evidence of interim progression between the completion of CNS- directed therapy and the screening radiographic study.
  6. Patients with new asymptomatic CNS metastases detected at the screening scan must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may then be eligible without the need for an additional brain scan prior to randomization, if all other criteria are met.
* Measurable disease, as defined by RECIST v1.1 Previously irradiated lesions can only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation and the previously irradiated lesion is not the only site of disease.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to randomization:

ANC ≥ 1500 cells/μL without granulocyte colony-stimulating factor support; Lymphocyte count ≥ 500/μL; Platelet count ≥ 100,000/μL without transfusion; Hemoglobin ≥ 9.0 g/dL; Patients may be transfused to meet this criterion. INR or aPTT ≤ 1.5 × upper limit of normal (ULN) This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose. AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN, with the following exceptions: Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN Patients with documented liver or bone metastases: alkaline phosphatase

* 5 × ULN. Serum bilirubin ≤ 1.25 × ULN Patients with known Gilbert disease who have serum bilirubin level ≤ 3 × ULN may be enrolled. Serum creatinine ≤ 1.5 × ULN

  * Patients must submit a pre-treatment tumor tissue sample during the study. Any available tumor tissue sample can be submitted. The tissue sample may be submitted after enrollment.
  * For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 90 days after the last dose of study treatment.

Exclusion Criteria:

* Active or untreated CNS metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 1 week prior to randomization
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Patients with indwelling catheters (e.g., PleurX®) are allowed.
* Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN) Patients who are receiving denosumab prior to randomization must be willing and eligible to discontinue its use and replace it with a bisphosphonate while in the study.
* Malignancies other than SCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous-cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
* Women who are pregnant, lactating, or intending to become pregnant during the study
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study. Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen are eligible for this study. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions: Rash must cover less than 10% of body surface area Disease is well controlled at baseline and only requires low potency topical steroids No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency, or oral steroids)
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Positive test for HIV
* Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to randomization. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
* Active tuberculosis
* Severe infections at the time of enrollment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Major surgical procedure other than for diagnosis within 28 days prior to randomization or anticipation of need for a major surgical procedure during the course of the study
* Prior allogeneic bone marrow transplantation or solid organ transplant
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk for treatment complications
* Previous anti-cancer therapy for ES-SCLC
* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 28 days prior to randomization
* Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation that such a live attenuated vaccine will be required during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multi-center study to compare the efficacy and safety of atezolizumab plus chemotherapy versus placebo plus chemotherapy in small cell lung cancer.
Sampling Method: Probability Sample
Enrollment: 1430 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 12 months
  Progression-free survival (PFS): refers to the time from the date of initiation of combination therapy to any objectively documented tumor progression or patient death (the last follow-up time for patients lost to follow-up; Patients who are still alive at the end of the study will be the end of follow-up at the end of the study).

SECONDARY OUTCOMES:
objective response rate | 12 months
  Objective response rate (ORR): refers to the proportion of patients whose tumors shrink to a certain amount and remain for a certain period of time, including complete response (CR) and partial response (PR) cases.
duration of response | 12 months
  Duration of response (DOR): refers to the duration of a patient's time from the first documented confirmed response (CR or PR) to the first documentation of disease progression (PD) or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No